CLINICAL TRIAL: NCT06924671
Title: GLA:D Back Canada - a Program for Persistent Low Back Pain.
Brief Title: GLA:D Back Canada - a Program for Chronic and Persistent Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00111890
Record Dates: First submitted 2025-04-05; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: GLA:D Back — GLA:D Back is a 10-week program based on first-line recommendations of patient education and structured exercise taught in a group format.

SUMMARY:
GLA:D Back is a program developed in Denmark to help people with persistent low back pain. This study will assist in contextualizing Danish content into an English version of the program.

DETAILED DESCRIPTION:
GLA:D Back is a program developed in Denmark to help people with persistent low back pain. Unfortunately, all materials developed for the program are in Danish. In this pilot, the investigators will translate the Danish materials into English, then use them to conduct an English training session for community clinicians in Edmonton, Alberta, Canada. Interested clinicians will then implement the program in their communities and provide feedback to contextualize the program for use in English. Specifically, surveys, interviews and focus groups will be used to help fine-tune the printed content of the course (e.g. manuals), it's training materials (e.g. lectures) and processes related to REDCap data collection (e.g. surveys).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent low back pain of at least 1 month's duration.

Exclusion Criteria:

* Participating currently in a supervised exercise or rehabilitation program or enrolled in another interventional clinical trial.
* Patients with nerve root involvement, suspected serious pathology, unstable trauma to the spine, aspects of pregnancy or other conditions that would prevent participation or disallow trial completion within the prescribed time period.
* Persons with conditions that require a specialist consult are suspected of needing a specialist consult, or have conditions that would be aggravated or worsened if treated by the interventions in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: English speaking adults greater than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Implementation | 6 months
  Number of clinicians who implement the program

SECONDARY OUTCOMES:
Patients enrolled | 6 months
  Number of patients trained by each GLA:D clinician

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No